CLINICAL TRIAL: NCT05032456
Title: Immersive Virtual Reality Improves Satisfaction In Laboring Women
Brief Title: Immersive Virtual Reality Satisfies the Women in Labor by Distracting Them From Their Labor Pain in Labor on Latent and Active Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Collaborators: Acibadem Maslak Hospital (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Dr. Selen Gür Özmen MD Phd, Assoc.Prof. Dr. Selen Gür Özmen, Bahçeşehir University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-18/07
Record Dates: First submitted 2021-07-20; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Labor Pain
Keywords: Labor; Immersive Virtual Reality; Non-pharmacologic Treatment; Anxiety; Depression
MeSH Terms: conditions — Labor Pain; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: 42 laboring women allocated to intervention group and control group randomly
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): Investigators used Oculus Quest All-in-one Virtual Reality Gaming Headset (128 GB) VR system. Before the intervention, the investigators introduced the equipment and instructed study participants on how to wear and activate the headsets. The laboring women who enrolled in the virtual reality group first wore the headsets in early labor (Cervical dilation 3 cm) for 20 minutes. The patients were offered to choose among several virtual environments including orange sunset, green meadows, black beginning, red savannah, blue deep, blue moon, blue ocean, white winter, and red fall. Cards printed out from the images of the Nature Trek application representing these novel immersion options were provided to the patients to help them pick up their preferred environment in advance. The second implementation of virtual reality headsets was after the epidural analgesia in the active phase of labor for another 20 minutes (Cervical dilation 6-7cm).
  Interventions: Device: Oculus Quest All-in-one VR Gaming Headset (128 GB) VR system
- Control Group (No Intervention): For participants randomized to the control group, virtual reality headsets were not used and the clinic's standard of care in laboring women was followed. Participants in this group filled out a visual pain rating scale both in the latent and active phases of labor.

INTERVENTIONS:
Device: Oculus Quest All-in-one VR Gaming Headset (128 GB) VR system — The laboring women who enrolled in the VR group were offered to choose among several virtual environments including orange sunset, green meadows, black beginning, red savannah, blue deep, blue moon, blue ocean, white winter, and red fall. Cards printed out from the screenshots of the Nature Trek application representing these novel immersion options were provided to the patients to help them pick up their preferred environment in advance.
  Arms: Virtual Reality Group

SUMMARY:
This is a randomized control study with 42 laboring women allocated to virtual reality intervention and control groups. The objective of this study, to evaluate the effectiveness of immersive virtual reality in laboring women on patient satisfaction and pain relief. The satisfaction of patients was measured with a "Virtual reality satisfaction survey" which was prepared by the investigators. Pain levels were assessed by a virtual pain rating scale in the early and the active phase of labor in both groups.

DETAILED DESCRIPTION:
Labor is a long and painful process for women. For avoiding or alleviating pain, adjuvant treatments such as hydrotherapy, yoga, hypnosis, acupuncture, and relaxation techniques could be used. Recent literature indicates the successful use of immersive virtual reality for a variety of painful medical procedures. Immersive virtual reality is hypothesized to reduce pain through distraction, a non-pharmacologic attentional mechanism. The user's brain is preoccupied with the flood of information presented by the virtual environment restricting the mind from processing pain signals. The investigators hypothesized that laboring women find immersive virtual reality as a beneficial tool for their overall labor and delivery experience. The 42 laboring women were randomized into two arms: virtual reality group ( intervention group) and control group. The investigators used Oculus Quest All-in-one VR Gaming Headset (128 GB) VR system. Before the intervention, the authors introduced the equipment and instructed study participants on how to wear and activate the headsets. Anxiety and depression scales were also applied on admission. The laboring women who enrolled in the VR group first wore the headsets in early labor (Cervical dilation 3 cm) for 20 minutes. The patients were offered to choose among several virtual environments including orange sunset, green meadows, black beginning, red savannah, blue deep, blue moon, blue ocean, white winter, and red fall. Cards printed out from the images of the Nature Trek application representing these novel immersion options were provided to the patients to help them pick up their preferred environment in advance. The second implementation of VR headsets was after the epidural analgesia in the active phase of labor for another 20 minutes (Cervical dilation 6-7cm). After the second intervention, the "Virtual Reality Satisfaction Survey" was applied by the authors. Patients were asked to fill out a visual pain rating scale right before and after the VR use in early and active labor. The primary objective of this study was to assessed whether immersive virtual reality provided pain relief in the latent or active phase of labor. The authors also evaluated anxiety and depression in both groups on admission as potential confounders. Anxiety and depression levels, assessed with the Beck Anxiety Inventory and Beck Depression Inventory. Patient satisfaction with the use of VR was assessed by a "Virtual Reality Satisfaction Survey" 10 question survey prepared by our team: 0 being the lowest and 100 being the highest possible VR satisfaction score.The investigators also asked these women whether the participants would like to use VR in future labor. Patient satisfaction with overall labor and delivery experience was assessed using a Visual Analog Scale (VAS). All discharged women were called a week following discharge and asked to rate their overall childbirth experience on a scale from 0 to 10. Zero indicates the most negative experience possible and 10 indicates the highest satisfaction possible. The authors classified a score of 8 to 10 as high satisfaction. Pain scores both in early and active labor in each group were assessed using Wong-Baker Faces Pain Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

* 18-42 years of age
* 37-41 week gestation
* A singleton pregnancy
* With vertex presentation
* No history of chronic medical conditions
* Absence of pregnancy complications
* Admission with documented labor by cervical exam and regular uterine contractions.

Exclusion Criteria:

* Migraine
* Headache
* Dizziness
* Motion Sickness
* Epilepsy
* Psychiatric disorders
* Visual or auditory disabilities
* History of cesarean section

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Being female and having singleton pregnancy at 37-41 weeks gestation
Enrollment: 42 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Virtual Reality Satisfaction Survey | During the intervention
  Patient satisfaction with the use of VR was assessed by a "Virtual Reality Satisfaction Survey" 10 question survey prepared by our team: 0 being the lowest and 100 being the highest possible VR satisfaction score.
Wong-Baker Faces Pain | During the intervention
  Pain scores both in early and active labor in each group were assessed using Wong-Baker Faces Pain Rating Scale. The scale shows a series of 6 faces ranging from a happy face at 0, or "no hurt", to a crying face at 5, which represents "hurts like the worst pain
Visual Analog Scale (VAS) | A week after the labor
  Patient satisfaction with overall labor and delivery experience was assessed using a Visual Analog Scale (VAS). Zero indicates the most negative experience possible and 10 indicates the highest satisfaction possible.

SECONDARY OUTCOMES:
Beck Anxiety Inventory (BAI) | Pre-intervention, on admission
  Anxiety levels of study participants were assessed with Beck Anxiety Inventory (BAI). [19] This inventory consists of 21 items, each scored from 0 to 3. This is a self-report questionnaire measuring somatic and cognitive parts of anxiety. The total score is calculated by finding the sum of 21 items. A score of 0 to 7 indicates minimal anxiety, 8 to 15 mild anxiety, 16 to 25 moderate anxiety, and 30 to 63 is associated with severe anxiety.
Beck Depression Inventory (BDI) | Pre-intervention, on admission
  It consists of 21 items which is a multiple-choice test and give a score ranging from 0 to 63. Each answer is scored on a scale value of 0-3. Measures of 0-9 indicate that a person is not depressed, 10-18 indicates mild-moderate depression, 19-29 indicates moderate-severe depression and 30-63 indicates severe depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem Maslak Hospital, Istanbul, Sariyer, Turkey (Türkiye)

REFERENCES:
- [Background] ACOG Committee Opinion #295: pain relief during labor. Obstet Gynecol. 2004 Jul;104(1):213. PMID 15229040
- [Background] Anim-Somuah M, Smyth RM, Cyna AM, Cuthbert A. Epidural versus non-epidural or no analgesia for pain management in labour. Cochrane Database Syst Rev. 2018 May 21;5(5):CD000331. doi: 10.1002/14651858.CD000331.pub4. PMID 29781504
- [Background] Nanji JA, Carvalho B. Pain management during labor and vaginal birth. Best Pract Res Clin Obstet Gynaecol. 2020 Aug;67:100-112. doi: 10.1016/j.bpobgyn.2020.03.002. Epub 2020 Mar 7. PMID 32265134
- [Background] Smith CA, Levett KM, Collins CT, Armour M, Dahlen HG, Suganuma M. Relaxation techniques for pain management in labour. Cochrane Database Syst Rev. 2018 Mar 28;3(3):CD009514. doi: 10.1002/14651858.CD009514.pub2. PMID 29589650
- [Background] Madden K, Middleton P, Cyna AM, Matthewson M, Jones L. Hypnosis for pain management during labour and childbirth. Cochrane Database Syst Rev. 2016 May 19;2016(5):CD009356. doi: 10.1002/14651858.CD009356.pub3. PMID 27192949
- [Background] Smith CA, Levett KM, Collins CT, Dahlen HG, Ee CC, Suganuma M. Massage, reflexology and other manual methods for pain management in labour. Cochrane Database Syst Rev. 2018 Mar 28;3(3):CD009290. doi: 10.1002/14651858.CD009290.pub3. PMID 29589380
- [Background] Dowswell T, Bedwell C, Lavender T, Neilson JP. Transcutaneous electrical nerve stimulation (TENS) for pain relief in labour. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD007214. doi: 10.1002/14651858.CD007214.pub2. PMID 19370680
- [Background] Maani CV, Hoffman HG, Morrow M, Maiers A, Gaylord K, McGhee LL, DeSocio PA. Virtual reality pain control during burn wound debridement of combat-related burn injuries using robot-like arm mounted VR goggles. J Trauma. 2011 Jul;71(1 Suppl):S125-30. doi: 10.1097/TA.0b013e31822192e2. PMID 21795888
- [Background] Mosadeghi S, Reid MW, Martinez B, Rosen BT, Spiegel BM. Feasibility of an Immersive Virtual Reality Intervention for Hospitalized Patients: An Observational Cohort Study. JMIR Ment Health. 2016 Jun 27;3(2):e28. doi: 10.2196/mental.5801. PMID 27349654
- [Background] Atzori B, Lauro Grotto R, Giugni A, Calabro M, Alhalabi W, Hoffman HG. Virtual Reality Analgesia for Pediatric Dental Patients. Front Psychol. 2018 Nov 23;9:2265. doi: 10.3389/fpsyg.2018.02265. eCollection 2018. PMID 30532720
- [Background] Walther-Larsen S, Petersen T, Friis SM, Aagaard G, Drivenes B, Opstrup P. Immersive Virtual Reality for Pediatric Procedural Pain: A Randomized Clinical Trial. Hosp Pediatr. 2019 Jul;9(7):501-507. doi: 10.1542/hpeds.2018-0249. Epub 2019 Jun 3. PMID 31160472
- [Background] Faruki A, Nguyen T, Proeschel S, Levy N, Yu J, Ip V, Mueller A, Banner-Goodspeed V, O'Gara B. Virtual reality as an adjunct to anesthesia in the operating room. Trials. 2019 Dec 27;20(1):782. doi: 10.1186/s13063-019-3922-2. PMID 31882015
- [Background] Wang YL, Gao HX, Wang JS, Wang JH, Bo L, Zhang TT, Dai YL, Gao LL, Liu Q, Zhang JJ, Cai JM, Yu JQ, Li YX. Immersive virtual reality as analgesia for women during hysterosalpingography: study protocol for a randomized controlled trial. Trials. 2020 Jan 20;21(1):102. doi: 10.1186/s13063-019-4023-y. PMID 31959220
- [Background] Hoffman HG, Richards TL, Coda B, Bills AR, Blough D, Richards AL, Sharar SR. Modulation of thermal pain-related brain activity with virtual reality: evidence from fMRI. Neuroreport. 2004 Jun 7;15(8):1245-8. doi: 10.1097/01.wnr.0000127826.73576.91. PMID 15167542
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Beck AT, Steer RA, Carbin MG. Psychometric properties of the Beck Depression Inventory: Twenty-five years of evaluation. Clinical Psychology Review. 1988.
- [Background] Shourab NJ, Zagami SE, Golmakhani N, Mazlom SR, Nahvi A, Pabarja F, Talebi M, Rizi SM. Virtual reality and anxiety in primiparous women during episiotomy repair. Iran J Nurs Midwifery Res. 2016 Sep-Oct;21(5):521-526. doi: 10.4103/1735-9066.193417. PMID 27904638
- [Background] Frey DP, Bauer ME, Bell CL, Low LK, Hassett AL, Cassidy RB, Boyer KD, Sharar SR. Virtual Reality Analgesia in Labor: The VRAIL Pilot Study-A Preliminary Randomized Controlled Trial Suggesting Benefit of Immersive Virtual Reality Analgesia in Unmedicated Laboring Women. Anesth Analg. 2019 Jun;128(6):e93-e96. doi: 10.1213/ANE.0000000000003649. PMID 31094789
- [Background] Kist M, Bekemeyer Z, Ralls L, Carvalho B, Rodriguez ST, Caruso TJ. Virtual reality successfully provides anxiolysis to laboring women undergoing epidural placement. J Clin Anesth. 2020 May;61:109635. doi: 10.1016/j.jclinane.2019.109635. Epub 2019 Oct 26. No abstract available. PMID 31662229
- [Background] Attanasio LB, McPherson ME, Kozhimannil KB. Positive childbirth experiences in U.S. hospitals: a mixed methods analysis. Matern Child Health J. 2014 Jul;18(5):1280-90. doi: 10.1007/s10995-013-1363-1. PMID 24072597
- [Background] Karlstrom A, Nystedt A, Hildingsson I. The meaning of a very positive birth experience: focus groups discussions with women. BMC Pregnancy Childbirth. 2015 Oct 9;15:251. doi: 10.1186/s12884-015-0683-0. PMID 26453022
- [Background] Dencker A, Bergqvist L, Berg M, Greenbrook JTV, Nilsson C, Lundgren I. Measuring women's experiences of decision-making and aspects of midwifery support: a confirmatory factor analysis of the revised Childbirth Experience Questionnaire. BMC Pregnancy Childbirth. 2020 Apr 6;20(1):199. doi: 10.1186/s12884-020-02869-0. PMID 32252679
- [Background] Tuncalp Ӧ, Were WM, MacLennan C, Oladapo OT, Gulmezoglu AM, Bahl R, Daelmans B, Mathai M, Say L, Kristensen F, Temmerman M, Bustreo F. Quality of care for pregnant women and newborns-the WHO vision. BJOG. 2015 Jul;122(8):1045-9. doi: 10.1111/1471-0528.13451. Epub 2015 May 1. No abstract available. PMID 25929823
- [Background] Lazzerini M, Mariani I, Semenzato C, Valente EP. Association between maternal satisfaction and other indicators of quality of care at childbirth: a cross-sectional study based on the WHO standards. BMJ Open. 2020 Sep 14;10(9):e037063. doi: 10.1136/bmjopen-2020-037063. PMID 32928854
- [Background] Jolles MW, de Vries M, Hollander MH, van Dillen J. Prevalence, characteristics, and satisfaction of women with a birth plan in The Netherlands. Birth. 2019 Dec;46(4):686-692. doi: 10.1111/birt.12451. Epub 2019 Sep 16. PMID 31524298
- [Background] Hawkins JL. Epidural analgesia for labor and delivery. N Engl J Med. 2010 Apr 22;362(16):1503-10. doi: 10.1056/NEJMct0909254. No abstract available. PMID 20410515
- [Background] Ashagrie HE, Fentie DY, Kassahun HG. A review article on epidural analgesia for labor pain management: A systematic review. International Journal of Surgery Open. 2020;24:100-4.
- [Background] Fyneface-Ogan S, Mato CN, Anya SE. Epidural anesthesia: views and outcomes of women in labor in a Nigerian hospital. Ann Afr Med. 2009 Oct-Dec;8(4):250-6. doi: 10.4103/1596-3519.59580. PMID 20139548
- [Background] Tulp MJ, Paech MJ. Analgesia for childbirth: modern insights into an age-old challenge and the quest for an ideal approach. Pain Manag. 2014 Jan;4(1):69-78. doi: 10.2217/pmt.13.63. PMID 24641345
- [Background] Lee SL, Liu CY, Lu YY, Gau ML. Efficacy of warm showers on labor pain and birth experiences during the first labor stage. J Obstet Gynecol Neonatal Nurs. 2013 Jan-Feb;42(1):19-28. doi: 10.1111/j.1552-6909.2012.01424.x. Epub 2012 Nov 20. PMID 23167574
- [Background] Gau ML, Chang CY, Tian SH, Lin KC. Effects of birth ball exercise on pain and self-efficacy during childbirth: a randomised controlled trial in Taiwan. Midwifery. 2011 Dec;27(6):e293-300. doi: 10.1016/j.midw.2011.02.004. Epub 2011 Apr 3. PMID 21459499
- [Background] Nieminen K, Stephansson O, Ryding EL. Women's fear of childbirth and preference for cesarean section--a cross-sectional study at various stages of pregnancy in Sweden. Acta Obstet Gynecol Scand. 2009;88(7):807-13. doi: 10.1080/00016340902998436. PMID 19488882
- [Background] Eyi EGY, Mollamahmutoglu L. An analysis of the high cesarean section rates in Turkey by Robson classification. J Matern Fetal Neonatal Med. 2021 Aug;34(16):2682-2692. doi: 10.1080/14767058.2019.1670806. Epub 2019 Oct 1. PMID 31570019
- [Derived] Carus EG, Albayrak N, Bildirici HM, Ozmen SG. Immersive virtual reality on childbirth experience for women: a randomized controlled trial. BMC Pregnancy Childbirth. 2022 Apr 23;22(1):354. doi: 10.1186/s12884-022-04598-y. PMID 35461248

DOCUMENTS (1):
  • Study Protocol (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT05032456/Prot_000.pdf